CLINICAL TRIAL: NCT01869361
Title: Randomized, Placebo Controlled Trial of Indomethacin for Tocolysis
Brief Title: Indomethacin for Tocolysis of Preterm Labor
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to much lower than expected numbers of eligible patients and lack of PI time, the study was not started.
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Kelly S Gibson, Maternal Fetal Medicine, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB13-00533
Record Dates: First submitted 2013-05-29; First posted 2013-06-05 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Preterm Labor
Keywords: preterm labor; tocolysis; indomethacin
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The patient will be given a loading dose of 50mg placebo by mouth followed by 25mg by mouth every six hours for a total of eight doses over 48 hours.
  Interventions: Drug: Placebo
- Indomethacin (Active Comparator): The patient will be given a loading dose of 50mg indomethacin by mouth followed by 25mg by mouth every six hours for a total of eight doses over 48 hours.
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Indomethacin — Study drug
  Other Names: Indocin
  Arms: Indomethacin
Drug: Placebo — Control drug
  Arms: Placebo

SUMMARY:
Indomethacin for tocolysis for 48 hours vs placebo

DETAILED DESCRIPTION:
Background: Indomethacin is frequently used as a tocolytic, however there is currently only scant evidence to support its efficacy.

Goals: To delay preterm delivery by 48 hours and to examine longer latency periods and maternal and neonatal outcomes Methods: Randomized placebo-controlled trial of indomethacin for tocolysis. Women with a singleton pregnancy between 23w0d and 31w6d in preterm labor randomly assigned to 50mg indomethacin by mouth followed by 25mg by mouth every 6hour for 48 hours or placebo. Patients receive betamethasone for fetal lung maturity, if not previously administered, and magnesium sulfate for neuroprotection. Ultrasound performed before initiation of study drug and after completion of study medication for amniotic fluid index and fetal cardiac assessment.

ELIGIBILITY:
Inclusion Criteria:

* Preterm labor as defined by regular uterine contractions (at least 6/hour) with cervical change of at least 1 cm or cervical shortening on transvaginal ultrasound less than 25mm of functional length
* Gestational age 23w0d to 31w6d weeks
* Singleton
* ≥ 18 years old
* Able to consent in English

Exclusion Criteria:

* Major congenital anomalies associated with an increased risk of newborn death
* Multiple fetal gestation (2+)
* Known intrauterine fetal demise
* Non-reassuring fetal status requiring delivery
* Preterm premature rupture of membranes (PPROM)
* Suspected or known intrauterine infection
* Placenta previa
* Maternal allergy or contraindication to indomethacin (peptic ulcer disease, thrombocytopenia, coagulopathy, renal or hepatic dysfunction)
* Inevitable delivery (cervix ≥6cm dilated)

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
delivery within 48 hours | 48 hours after enrollment
  The percentage of patients remaining undelivered after 48 hours

SECONDARY OUTCOMES:
delivery within 7 days | 7 days after enrollment
  The percentage of patients remaining undelivered after 7 days
delivery before 37 weeks | participants will be followed for the duration of pregnancy through their postpartum period, an expected time of up to 20 weeks
  The percentage of patients remaining undelivered until 37 weeks gestational age
Maternal and Fetal Complications | participants will be followed for the duration of pregnancy through their postpartum period and neonatal hospital stay, an expected time of up to 24 weeks
  composite of maternal intolerance of the drug, birth weight, gestational age, neonatal morbidities, changes in amniotic fluid volume, fetal cardiac assessment, or premature constriction of the ductus arteriosus.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly S Gibson, MD, Principal Investigator — MetroHealth Medical Center; Brian Mercer, MD, Study Chair — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists; Committee on Practice Bulletins-Obstetrics. ACOG practice bulletin no. 127: Management of preterm labor. Obstet Gynecol. 2012 Jun;119(6):1308-17. doi: 10.1097/AOG.0b013e31825af2f0. PMID 22617615
- [Background] Haas DM, Caldwell DM, Kirkpatrick P, McIntosh JJ, Welton NJ. Tocolytic therapy for preterm delivery: systematic review and network meta-analysis. BMJ. 2012 Oct 9;345:e6226. doi: 10.1136/bmj.e6226. PMID 23048010
- [Background] Hayes E, Moroz L, Pizzi L, Baxter J. A cost decision analysis of 4 tocolytic drugs. Am J Obstet Gynecol. 2007 Oct;197(4):383.e1-6. doi: 10.1016/j.ajog.2007.06.052. PMID 17904969
- [Background] Abramovici A, Cantu J, Jenkins SM. Tocolytic therapy for acute preterm labor. Obstet Gynecol Clin North Am. 2012 Mar;39(1):77-87. doi: 10.1016/j.ogc.2011.12.003. Epub 2012 Jan 4. PMID 22370109
- [Background] Zuckerman H, Shalev E, Gilad G, Katzuni E. Further study of the inhibition of premature labor by indomethacin. Part II double-blind study. J Perinat Med. 1984;12(1):25-9. doi: 10.1515/jpme.1984.12.1.25. PMID 6374098
- [Background] Niebyl JR, Blake DA, White RD, Kumor KM, Dubin NH, Robinson JC, Egner PG. The inhibition of premature labor with indomethacin. Am J Obstet Gynecol. 1980 Apr 15;136(8):1014-9. doi: 10.1016/0002-9378(80)90629-8. PMID 7369252
- [Background] Panter KR, Hannah ME, Amankwah KS, Ohlsson A, Jefferies AL, Farine D. The effect of indomethacin tocolysis in preterm labour on perinatal outcome: a randomised placebo-controlled trial. Br J Obstet Gynaecol. 1999 May;106(5):467-73. doi: 10.1111/j.1471-0528.1999.tb08300.x. PMID 10430197
- [Background] Amin SB, Sinkin RA, Glantz JC. Metaanalysis of the effect of antenatal indomethacin on neonatal outcomes. Am J Obstet Gynecol. 2007 Nov;197(5):486.e1-10. doi: 10.1016/j.ajog.2007.04.019. PMID 17980183
- [Background] Sood BG, Lulic-Botica M, Holzhausen KA, Pruder S, Kellogg H, Salari V, Thomas R. The risk of necrotizing enterocolitis after indomethacin tocolysis. Pediatrics. 2011 Jul;128(1):e54-62. doi: 10.1542/peds.2011-0265. Epub 2011 Jun 20. PMID 21690109
- [Background] Loe SM, Sanchez-Ramos L, Kaunitz AM. Assessing the neonatal safety of indomethacin tocolysis: a systematic review with meta-analysis. Obstet Gynecol. 2005 Jul;106(1):173-9. doi: 10.1097/01.AOG.0000168622.56478.df. PMID 15994634
- [Background] Cordero L, Nankervis CA, Gardner D, Giannone PJ. The effects of indomethacin tocolysis on the postnatal response of the ductus arteriosus to indomethacin in extremely low birth weight infants. J Perinatol. 2007 Jan;27(1):22-7. doi: 10.1038/sj.jp.7211612. Epub 2006 Oct 19. PMID 17053778
- [Background] Eronen M, Pesonen E, Kurki T, Ylikorkala O, Hallman M. The effects of indomethacin and a beta-sympathomimetic agent on the fetal ductus arteriosus during treatment of premature labor: a randomized double-blind study. Am J Obstet Gynecol. 1991 Jan;164(1 Pt 1):141-6. doi: 10.1016/0002-9378(91)90644-7. PMID 1986601
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046